CLINICAL TRIAL: NCT00785122
Title: An Open Label, Multicenter Phase 1-2 Study to Investigate the Effectiveness, Safety and Immunogenicity of a Monotherapy With Intradermal IMA910 Plus GM-CSF Following Pre-treatment With Low-dose Cyclophosphamide in Advanced Colorectal Carcinoma Patients Who Have Successfully Completed a 12 Week First-line Treatment With Oxaliplatin-based Chemotherapy.
Brief Title: IMA910 Plus GM-CSF With Low-dose Cyclophosphamide Pre-treatment in Advanced Colorectal Carcinoma Patients Following a Successful 12 Week First-line Treatment With Oxaliplatin-based Chemotherapy (IMA910-101)
Acronym: IMA910-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immatics Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT Nr. 2007-005666-12
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Carcinoma
Keywords: cancer vaccine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sargramostim; Cyclophosphamide; Imiquimod; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Endoxana, Leukine, IMA910 — a single i.v. infusion of 300 mg/m2 Endoxana (Cyclophosphamide) and then 3 days later (visit 1) patients will start vaccination therapy with intradermal (i.d.) injections of 75µg GM-CSF followed by i.d. injections of 5.78 mg IMA90
  Other Names: Endoxana (Cyclophosphamide); Aldara (Imiquimod); IMA910; GM-CSF
Drug: Endoxana, Leukine, IMA910, Aldara — a single i.v. infusion of 300 mg/m2 Endoxana (Cyclophosphamide) and then 3 days later (visit 1) patients will start vaccination therapy with intradermal (i.d.) injections of 75µg GM-CSF followed by i.d. injections of 5.78 mg IMA90 followed by Aldara (Imiquimod)
  Other Names: Endoxana (Cyclophosphamide); Aldara (Imiquimod); IMA910; GM-CSF

SUMMARY:
This study is being conducted in order determine whether IMA910 as single agent with GM-CSF as adjuvant following pre-treatment with low-dose cyclophosphamide is safe and shows sufficient anti-tumour effectiveness in patients with advanced CRC to warrant further development. Secondary objectives of this study are investigation of immunological parameters and additional effectiveness endpoints. Furthermore, safety, immunological parameters and effectiveness of IMA910 as single agent with GM-CSF in combination with imiquimod following pre-treatment with low-dose cyclophosphamide will be investigated in a 2nd cohort of patients.

The regular study duration for individual patients in the 1st and 2nd cohort comprises regularly 18-42 days of screening (excluding HLA-typing), 33 weeks of treatment (16 vaccinations) and 4 weeks follow-up. Thus, the period between start of screening and end of trial is about 10 months per patient. Patients will be followed for response to subsequent treatments (chemotherapies with or without targeted agents) and survival every 2 months after EOS visit until death.

Patients in the 1st and 2nd cohort will be withdrawn from study treatment once a progress according to RECIST is noted. An enrolment plan for the first 6 patients included into the 1st cohort will be part of this study to ensure maximum safety of the study participants. The enrollment of the first 6 patients into the 2nd cohort will also follow an enrolment plan to ensure maximum safety.

DETAILED DESCRIPTION:
This is a multicentre, open-label, Phase 1-2 study in patients with locally advanced and/or metastatic colorectal cancer (CRC) to investigate the effectiveness, safety and immunogenicity of the tumour multi-peptide vaccine IMA910 plus GM-CSF (1st cohort) given as monotherapy after successful (CR, PR or SD) completion of a 12 week first-line oxaliplatin-based standard chemotherapy (e.g. FOLFOX, XELOX). Safety, immunogenicity and effectiveness of IMA910 plus GM-CSF in combination with imiquimod will be investigated in a 2nd cohort of patients with locally advanced and/or metastatic colorectal cancer (CRC) after successful (CR, PR or SD) completion of a 12 week first-line oxaliplatin-based standard chemotherapy (e.g. FOLFOX, XELOX).

The aim of this study is to investigate whether IMA910 plus GM-CSF (1st cohort) is an effective maintenance therapy with a favorable toxicity profile. A single dose of low-dose cyclophosphamide is applied as an immune modulator 3 days before the start of vaccination. Effectiveness is measured in terms of the disease control rate (DCR) at Visit 14 (= 27 weeks of vaccination) according to RECIST. The baseline tumour response assessment is performed after a first-line oxaliplatin-based standard chemotherapy for 12 weeks. The DCR is compared to a no effect level of 21% derived from the PFS curve of the chemotherapy-free interval cohort (arm B) of the OPTIMOX 2 study. Tumour response assessments will be performed every 9 weeks according to RECIST. Further a 2nd cohort of patients will be treated with IMA910 plus GM-CSF in combination with imiquimod and a single dose of lowdose cyclophosphamide. The aim of the 2nd cohort is to investigate whether the addition of imiquimod is safe, enhances the immune response to IMA910 and shows effectiveness.

Patients in the 1st and 2nd cohort will be withdrawn from study treatment once a progress according to RECIST is noted. An enrolment plan for the first 6 patients included into the 1st cohort will be part of this study to ensure maximum safety of the study participants. The enrollment of the first 6 patients into the 2nd cohort will also follow an enrolment plan to ensure maximum safety.

Patients must be HLA-A*02-positive. Patients must have been diagnosed with unresectable, locally advanced and/or metastatic colorectal cancer before first-line chemotherapy. Patients must have completed a 12 week first-line oxaliplatin-based standard chemotherapy (e.g. FOLFOX or XELOX) with either complete or partial response or stable disease as the outcome. In case the 12 week first-line oxaliplatin-based standard chemotherapy results in resectable disease the patient may not be enrolled and routinely undergoes surgical resection of residual tumour. Patients must be aged 18 years or older and must have histological confirmed colorectal adenocarcinoma (CRC) and radiological evidence (CT/MRI) of unresectable locally advanced and/or metastatic CRC prior to 12 week first-line oxaliplatin-based standard chemotherapy.

This study will employ low-dose Cyclophosphamide (administered as a single i.v. infusion at a dose of 300 mg/m2 3 days prior to the vaccination) in order to increase the immune response to IMA910 (5.78 mg i.d.). Patients will receive 7 vaccinations of IMA910 plus GM-CSF (75 μg i.d.) in the first 6 weeks of treatment (induction period) followed by 9 vaccinations at 3-week intervals for a further 27 weeks (maintenance period). The patients will receive a total of 16 vaccinations over a period of 33 weeks. An end of study visit (EOS, Visit 17) will be performed 4 weeks after the last treatment. Patients enrolled into the 2nd cohort of the study will receive the same treatment as described above and will additionally receive a topical application of 250 mg imiquimod cream (12.5 mg imiquimod) 10 minutes (up to 20 minutes) after each application of IMA910 (Visit 1-16) and from day 3 onwards 250 mg imiquimod cream (12.5 mg imiquimod) 24 hours (but up to 48 hours at the latest) after each application of IMA910 (Visit 3-16). The topical application of imiquimod additionally 24 hours (but up to 48 hours at the latest) after IMA910 application will be done by the patient at home. Imiquimod cream will be applied to a marked 5x5 cm area around the injection site of GM-CSF and IMA910.

At screening a CT or MRI of the chest and abdomen/pelvis will be performed to assess baseline tumour status. In patients with suspected brain metastasis at Screening or if clinically indicated a CT or MRI of the brain will be performed. In patients with known bone metastases of the extremities or in case of suspected bone metastases of the extremities at Screening correlative imaging (X-ray, CT or MRI) has to be performed of the respective area(s). At Visits 8, 11, 14, and 17 (EOS) a CT or MRI of the chest, abdomen and pelvis will be performed. In patients with bone metastases of the extremities detected at baseline or during the study, repeat assessments of the sites of bone metastases (X-ray, CT or MRI) will be performed at Visits 14 and 17 (EOS). An assessment of brain metastasis will be performed only if clinically indicated during the course of the study.

Cellular immunomonitoring (T-cell responses to peptides contained in IMA910 and analysis of other immune cell populations that may influence T-cell responses such as Tregs), serum levels of antibodies and molecules with suspected influence on immune response will be assessed on several occasions during the study. In a subgroup of patients the following parameters may be assessed in tumour tissue (depending on the amount and quality of tissue): expression of target genes encoding the TUMAPs contained in IMA910 and of genes which might be influenced by IMA910, presentation of TUMAPs contained in IMA910, presence of tumour infiltrating lymphocytes and presence of molecules with suspected influence on immune response.

Safety assessment will comprise continuous adverse event reporting, regular physical examinations and regular assessments of vital signs, haematology, blood chemistry and urine. A 12-lead ECG will be performed at screening and at the end of the study. Pregnancy testing will be performed according to applicable legislation in the country where the trial is being performed. At the very least, women of childbearing potential must undergo a pregnancy test during screening for the study, before the first dose and at the end of the study.

In the initial phase of the study 6 patients of the 1st Cohort will be treated step-wise and observed for 21 days according to a pre-specified enrolment plan. The first step is the enrolment of 1 patient followed by an observation period of 21 days, thereafter enrolment of 2 patients followed by an observation period of 21 days thereafter 3 patients followed by an observation period of 21 days. The sponsor will evaluate the adverse events and laboratory data following every enrolment step and initiate the enrolment of the next enrolment step. After 6 patients enrolled in that way the subsequent enrolment can be performed without further restrictions.

Further also in the 2nd Cohort the first 6 patients of the 2nd cohort will be enrolled in a step-wise manner. The first step is the enrolment of 1 patient followed by an observation period of 1 week, thereafter enrolment of 2 patients followed by an observation period of 1 week thereafter enrolment of 3 patients followed by an observation period of 1 week. The sponsor will evaluate the adverse events following every enrolment step and initiate the enrolment of the next enrolment step. After 6 patients enrolled in that way the subsequent enrolment can be performed without further restrictions.

ELIGIBILITY:
Inclusion criteria:

* Aged at least 18 years
* HLA type: HLA-A*02-positive
* Histologically confirmed colorectal adenocarcinoma (CRC)
* Radiological evidence (CT/MRI) of unresectable locally advanced and/or metastatic CRC prior to 12 week first-line oxaliplatin-based standard chemotherapy
* 12 week first-line chemotherapy with an oxaliplatin-based regimen according to an established standard protocol (e.g. FOLFOX or XELOX) administered at the following minimum dosages over this 12 week period: Oxaliplatin 400 mg/m2, Fluorouracil (5FU) 10.000 mg/m2 or Capecitabine 84.000 mg/m2 (a time window for application of first-line chemotherapy of +4 weeks is allowed)
* Response (CR, PR) or stabilization (SD) following a 12 week first-line oxaliplatin-based standard chemotherapy shown by radiological evidence (CT/MRI after last cycle of firstline oxaliplatin-based standard chemotherapy compared to CT/MRI taken before start of first-line oxaliplatin-based standard chemotherapy)
* Patients accept a chemotherapy-free interval under close observation (CT or MRI scans performed every 9 weeks)
* Maximum period between start of study treatment (Cyclophosphamide) and start of the last cycle of standard chemotherapy (= first day of last cycle of standard chemotherapy) is 42 days; minimum period is 18 days
* Karnofsky Performance Status ≥80%
* Able to understand the nature of the study and give written informed consent
* Willing and ability to comply with the study protocol for the duration of the study

Exclusion criteria:

* Any adjuvant systemic or local chemotherapy if ended ≤6 months before start of systemic first-line oxaliplatin-based standard chemotherapy
* Progressive disease during or at the end of 12 week systemic first-line oxaliplatin-based standard chemotherapy
* CT/MRI scans taken more than 9 weeks before start of first-line oxaliplatin-based standard chemotherapy
* Response to 12 week first-line oxaliplatin-based standard chemotherapy resulting in resectable disease; curative treatment intended
* Immunosuppressive therapy within 10 days before first vaccination e.g. corticosteroid treatment (inhalative corticosteroids for e.g. asthma are allowed)
* Radiotherapy during and/or following the 12 week first-line oxaliplatin-based standard chemotherapy (palliative radiotherapy for bone metastasis is allowed)
* Concurrent or prior participation in a clinical trial applying interventional procedures (e.g. application of investigational drugs, surgical interventions) within the last 30 days before Screening 2 = Visit B
* History of other malignant tumours within the last 5 years, except basal cell carcinoma or curatively excised cervical carcinoma in situ
* Presence of known brain metastasis on MRI or CT scans
* Current partial or complete bowel obstruction
* Patients with a history or evidence of systemic autoimmune disease
* Any vaccination within 2 weeks before first vaccination
* Any planned prophylactic vaccination from study entry until the end of the induction period (Week 6 after first vaccination, exception: if medically indicated)
* Major surgery ≤4 weeks before first vaccination
* Any of the following abnormal laboratory values:

  * Haematology:

    * Hb <9 g/dL
    * WBC <2.5 x 109/L
    * Neutrophils <1.5 x 109/L
    * Lymphocytes <1.0 x 109/L
    * Platelets <75 x 109/L
  * Liver function:

    * Serum bilirubin >1.5 x upper normal limit (unless a history of Gilbert's disease)
    * ALAT or ASAT >3 x upper normal limit (>5 x ULN if liver metastases are present)
    * Alkaline Phosphatase >3 x upper normal limit (>5 x ULN if liver metastases are present)
  * Renal function: serum creatinine >200 μmol/L (2.3 mg/dL)
* Known active hepatitis B or C infection
* Known HIV infection
* Active infections requiring oral or intravenous antibiotics
* Any other infection with a biological agent that can cause a severe disease and poses a severe danger to lab personnel working on patient tissues. Examples are: rabies, Mycobacterium tuberculosis, Coccidioides immitis
* Patients with other significant diseases currently uncontrolled by treatment which might interfere with study completion, including gastrointestinal, hepatic, renal, respiratory, cardiovascular, haematological, coagulation, metabolic or hormonal diseases with clinically relevant abnormal organ function for example:

  * Heart failure or non-compensated active heart disease (=NYHA Class III and IV)
  * Severe coronary heart disease, cardiac arrhythmia requiring medication, or uncontrolled hypertension
  * Symptomatic neurotoxicity (motor or sensory) = Grade 3 according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE)
  * Severe pulmonary dysfunction
* Psychiatric disabilities, seizures or central nervous system disorders that may interfere with the ability to give informed consent or perform adequate follow-up in the investigator's opinion
* Pregnancy or breast-feeding
* Hypersensitivity to the study drugs (cyclophosphamide, GM-CSF, IMA910) including excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Disease control rate | after 27 weeks of vaccination
Safety assessment | continuously
  Safety assessment with special emphasis on the inclusion of the first 6 patients enrolled according to a pre-specified enrolment plan

SECONDARY OUTCOMES:
Tumour response rates and SD rate | after 27 and 37 weeks
DCR | after 37 weeks on study
Duration of response | till End of Study
Progression free survival | until tumor progression or death
Cellular immunomonitoring | till 27 weeks of vaccination or End Of Study
  * T-cell responses to peptides contained in IMA910
  * Description of T-cell responses
  * Percentage of multipeptide responders
  * Number of TUMAPs to which a response can be detected in multipeptide responders
  * Other immune cell populations that may influence T-cell responses such as regulatory T cells
Biomarkers | Pre-Vaccination and End of Study
  Pre-vaccination and post-vaccination analysis of serum markers with suspected influence on success of vaccination such as cytokines.
Analysis of tumor tissue | optional if available
  Depending on the amount, type & quality parameters may be assessed:
  * Analysis of expression of tumor genes influencing immune response
  * Presentation of TUMAPs contained in IMA910
  * Tumor infiltrating lymphocytes and other immune cell populations
  * Presence of molecules with suspected influence on immune response
  * Alteration in the tumor signature under the influence of study treatment with respect to expression of the target genes encoding the TUMAPs contained in IMA910 and all the above mentioned parameters
Overall Safety | continuously till End of Study
Effect of imiquimod (2nd Cohort) on immune response | till End of Study
  All effectiveness and immunological endpoints will be analysed separately for the
  1st and the 2nd cohort. Overall safety, biomarkers and analysis of tumour tissue will be analysed separately for the 1st and the 2nd cohort and additionally overall for both cohorts.
Overall survival | unitl death
Non-Cellular immunomonitoring | till 27 weeks of vaccination
  * Serum levels of antibodies directed against peptides contained in IMA910 and against MHC/peptide complexes thereof
  * Presence of molecules with suspected influence on immune response such as serum TGFβ

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Mayer-Mokler, Study Director — immatics biotechnolgies GmbH
Locations (41):
- Belgium (2):
  - Medische Oncologie, Imeldaziekenhuis, Bonheiden
  - Oncologisch Centrum, UZ Gent, Ghent
- Bulgaria (5):
  - Inter District Dispencary for Oncology Disease with Inpatient Unit Plovdiv, First Internal Ward, Plovdiv
  - District Dispensary for Oncology Diseases with Inpatient Unit, Sofia District, Chemotherapeutic Ward, Sofia
  - MHAT "Tsaritsa Yoanna", Clinic of Oncotherapy, Sofia
  - Specialized Hospital for Active Treatment in Oncology Ltd., Clinic of Chemotherapy, Sofia
  - Interdistrict Dispensary of Oncology Diseases with Inpatient Unit "Dr. Marko Markov" - Varna, Varna
- Germany (7):
  - University Hospital Dresden "Carl Gustav Carus", Dresden
  - Krankenhaus Nordwest der Stiftung Hospital zum heiligen Geist, II. med. Klinik, Frankfurt a.M.
  - Cancer Hospital Sanafontis, Freiburg im Breisgau
  - Prosper-Hospital, Med. Klinik I, Recklinghausen
  - University of Tübingen, Department of med. Oncology, Hematology, Immunology, Rhematology and Pulmology, Tübingen
  - Universitätsklinikum Ulm, Dep. Of Internal Medicine I, Studiensekretariat, CCCU, CTOA, Ulm
  - Kliniken Villingen, Schwarzwald-Baar-Klinik, Dept. Of Hematology & Oncology, Villingen-Schwenningen
- Hungary (8):
  - State Health Center Oncology, Budapest
  - Péterfy Hospital, Budapest
  - Semmelweis University, Oncoradiology, Budapest
  - National Institute of Oncology, Department of Internal Medicine, Department of Chemotherapy "B", Budapest
  - Uszoki Hospital, Budapest
  - Borsod County Hospital, Miskolc
  - University of Szeged, Department of Oncotherapy, Szeged
  - St. Gyorgy County Hospital, Székesfehérvár
- Latvia (2):
  - Pauls Stradins University Hospital, Riga
  - Latvia oncological Center, Riga
- Poland (4):
  - Centrum Onkologii Instytut im. Marii Skłodowskiej-Curie Klinika Onkologii Klinicznej, Gliwice
  - Klinika Chemioterapii Nowotworów, Regionalny Ośrodek Onkologiczny, Wojewódzki Szpital Specjalistyczny im. M.Kopernika Uniwersytetu Medycznego Łódz, Lodz
  - Wojewodzki Szpital Zespolony im. Ludwika Rydygiera, Oddzial Chemiotherapii, Torun
  - Katedra i Klinika Hematologii, Onkologii i Cherob Wewnetrznych AM SP Centralny Szpital Kliniczny w Warszawie, Warsaw
- Romania (3):
  - Oncology Institute "Prof. Dr. Ion Chiricuta", Cluj-Napoca
  - Clinical County Hospital Oradea, Oncology Clinic, Oradea
  - Spitalul Clinic Judetean, Târgu Mureş
- Serbia (3):
  - Institute for Oncology and Radiology of Serbia, National Cancer Research Center, Clinical Research and Exp. Pharmacology, Belgrade
  - Vojnomedicinska Akademija, Clinic for Gastroenterology, Military Medical Academy, Belgrade
  - Oncology Institute of Vojvodina, Sremska
- United Kingdom (7):
  - The Royal Sussex County Hospital, CIR-Unit, Brighton
  - University of Cambridge, Department of Oncology, Cambridge
  - Velindre Cancer Centre, Cardiff
  - St Luke's Cancer Centre, The Royal Surrey County Hospital, Guildford / Surrey
  - St. James's Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Churchill Hospital, Dept.of Clinical Pharmacology, Oxford